CLINICAL TRIAL: NCT03402139
Title: Molecular Basis of Early Childhood Obesity Programming by Intrauterine Growth Restriction
Brief Title: Early Childhood Obesity Programming by Intrauterine Growth Restriction
Status: Recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Icahn School of Medicine at Mount Sinai (Other); Hackensack Meridian Health Center for Discovery and Innovation (Unknown); University of California, San Francisco (Other); University of Wisconsin, Madison (Other); Gencove (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-8749; R01HD092533 (NIH)
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Childhood Obesity; Epigenetics
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will collect cord and peripheral blood, buccal swab, urine and stool samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IUGR infants: Intrauterine growth restricted infants will be enrolled. There are no interventions.
- AGA infants: Appropriate for gestational age infants will be enrolled. There are no interventions.

SUMMARY:
The molecular mechanisms underlying developmental programming of childhood obesity remain poorly understood. Here, the investigators address major questions about early childhood obesity programming by studying CD3+ T-cells from intrauterine growth restricted (IUGR) newborns who have an increased risk for obesity and other metabolic disorders in adult life.

DETAILED DESCRIPTION:
Epidemiological studies of multiple cohorts suggest an increased risk for obesity, cardiovascular disease-related death and type 2 diabetes in low birth weight infants. However, the molecular mechanisms underlying developmental programming of childhood obesity remain poorly understood. Alterations in DNA methylation during fetal life have been proposed to be one of the mechanisms that regulate this phenotype. Here, the investigators address major questions about early childhood obesity programming by studying purified subpopulations of CD3+ T-cells from intrauterine growth restricted (IUGR) newborns who have an increased risk for obesity and other metabolic disorders in adult life. The investigators will correlate altered CD3+ T-cell DNA methylation profiles in cord and peripheral blood samples and functional changes in CD3+ T-cells with adiposity in childhood.

ELIGIBILITY:
Mother-infant pairs will be recruited for this study.

Inclusion Criteria:

* Healthy singleton term intrauterine growth restricted (IUGR) and appropriate for gestational age (AGA) infants whose mothers are followed by the Obstetric Department of Montefiore Medical Center and who deliver at the Weiler Division of Montefiore Medical Center. Infants will be classified as IUGR if birth weight is <10th percentile for gestational age and gender based on World Health Organization (WHO) growth curves. Infants will be classified as AGA if birth weight percentile is >10th and <90th percentile
* Reproductive age women, healthy enough to achieve pregnancy
* Deliver a single healthy live term infant at ≥37 weeks' gestational age (GA)
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Multiple gestation
* Maternal depression
* Maternal renal disease
* History of maternal smoking in the 2nd and 3rd trimester of pregnancy
* Maternal gestational diabetes / Type 2 Diabetes (T2D)
* Preterm birth (less than 37 weeks' gestation)
* Known chromosomal or congenital anomaly
* Infants in extremis
* Low Apgar scores (Apgar score <7 at 5 minutes of age)
* Known congenital bacterial or non-bacterial infections
* Known inborn errors of metabolism

Ages: 1 Hour to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term AGA and IUGR singleton infants
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Growth velocity | Until 24 months of age
  Change in growth velocity based on DNA methylation marks and functional profiles of CD3+ T-cells
DNA methylation of CD3+ T-cells | At birth and 24 months of age
  Change in DNA methylation of CD3+ T-cells in the first 24 months of life in IUGR infants
T-cell function | At birth, 12 and 24 months of age
  Change in T-cell function in the first 24 months of life in IUGR infants

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Reznik, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Jack D. Weiler Hospital, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No